CLINICAL TRIAL: NCT07036614
Title: The Application of Novel Special Light in the Diagnosis of Endotracheal/Bronchial Lesions.
Brief Title: The Novel Special Light for Endotracheal/Bronchial Lesions.
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Other Study IDs: SHCHE202409
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-01

CONDITIONS: Tracheal Disease; Bronchial Disease
Keywords: TXI; NBI; RDI; WLI
MeSH Terms: conditions — Tracheal Diseases; Bronchial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with endotracheal/bronchial lesions.: Approximately 400 patients who meet the inclusion and exclusion criteria will be enrolled to develop and validate the the Novel Special Light for the diagnosis of endotracheal/bronchial lesions.

SUMMARY:
This is a single-center study. The purpose of this study is o evaluate the diagnostic value of special light (TXI, NBI, RDI) in endotracheal/bronchial lesions.

DETAILED DESCRIPTION:
The latest endoscopic system, EVIS X1 (Olympus Medical Systems, Tokyo, Japan), was developed in 2020, which includes brighter and clearer WLI, third-generation (3G)-NBI, texture and color enhancement imaging (TXI) ,and red dichromatic imaging (RDI) as a new image-enhanced endoscopy (IEE) . texture and color enhancement imaging (TXI) as a new image-enhanced endoscopy (IEE). The TXI is designed to enhance the 3 image elements of WLI (texture, brightness, and color) using Retinex-based enhancements while maintaining image naturalness (WLI appearance) clearly defines subtle tissue differences. RDI enables observation of deeper tissue regions by utilizing light of longer wavelengths; such light has weak light scattering characteristics, thus providing the opposite effect of NBI. The original purpose of RDI was to reduce the risk of bleeding during endoscopic treatment by improving the visibility of thick blood vessels in deeper tissues. Although great efforts have been made in exploring the various clinical efficacies of RDI, no published reports have comprehensively covered both the technological and clinical aspects of RDI. The purpose of this study is o evaluate the diagnostic value of special light (TXI, NBI, RDI) in endotracheal/bronchial lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Patients with chest imaging findings indicating central lung lesions requiring further bronchoscopy;
3. Patients with neoplasm in the lumen that could be biopsied by bronchoscopy or operated;
4. Patient who has good compliance and sign informed consent;
5. The investigator believes that the subjects can understand the process of the clinical study, are willing and able to complete all the research procedures and follow-up visits, and cooperate with the research procedures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. No endotracheal/bronchial lesions were detected by bronchoscopy;
3. Allergic reaction to narcotic drugs in previous medical history;
4. The investigator believes that the subject is not suitable for bronchoscopy;
5. High-risk diseases or other special conditions for which the investigator considers the subjects unsuitable for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endotracheal/bronchial lesions scheduled for a bronschoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the special light for endotracheal/bronchial Lesions. | 1month
  Histopathology will be used as the gold standard. To compare the diagnostic value of the special light (TXI, NBI, RDI) and white light (WLI) in differential diagnosis of benign and malignant luminal lesions.

SECONDARY OUTCOMES:
The diagnostic methods and grading criteria of the special light | 1 month
  Based on the special light (TXI, NBI, RDI), the diagnostic methods and grading criteria for benign and malignant endotracheal/bronchial lesions were established.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may release the database after the study, but no decision has been made yet.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342